CLINICAL TRIAL: NCT00744861
Title: EXO-SPINE: A Prospective, Multi-center, Double-blind, Randomized, Placebo Controlled Pivotal Study of Ultrasound as Adjunctive Therapy for Increasing Posterolateral Fusion Success Following Single Level Posterior Instrumented Lumbar Surgery
Brief Title: Ultrasound as Adjunct Therapy for Increasing Fusion Success After Lumbar Surgery
Acronym: EXO-SPINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated following interim analysis
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-SPINE0907
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Lumbar Degenerative Disc Disease
Keywords: Lumbar Fusion; exospine; Exo-Spine; LIPUS; Exogen
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exogen 4000+ (Active Comparator): Low intensity pulsed ultrasound (LIPUS) delivered via Exogen 4000+ (single transducer) device for a treatment duration of 20 minutes per fusion site per day.
  Interventions: Device: Exogen 4000+
- Exogen 4000+ sham (Sham Comparator): Non-active sham device identical to Exogen 4000+ (single transducer); treatment duration of 20 minutes per fusion site per day
  Interventions: Device: Exogen 4000+ sham
- Exospine (Active Comparator): Low intensity pulsed ultrasound delivered via Exospine device (dual transducers); treatment duration of 20 minutes per day
  Interventions: Device: Exospine
- Exospine sham (Sham Comparator): Non-active sham device identical to Exospine (dual transducers); treatment duration of 20 minutes per day
  Interventions: Device: Exospine sham

INTERVENTIONS:
Device: Exospine sham — Inactive Exospine LIPUS device (dual transducers)
  Arms: Exospine sham
Device: Exospine — Active Exospine LIPUS device (dual transducers)
  Arms: Exospine
Device: Exogen 4000+ — Active Exogen LIPUS device (single transducer)
  Arms: Exogen 4000+
Device: Exogen 4000+ sham — Inactive Exogen 4000+ LIPUS device (single transducer)
  Arms: Exogen 4000+ sham

SUMMARY:
Adjunct therapy for increasing posterolateral fusion success following single level posterior instrumented lumbar surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether using active low intensity pulsed ultrasound as adjunct therapy following single level posterior instrumented lumbar surgery increases the posterolateral success rate when compared to inactive (placebo) therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a documented diagnosis of degenerative disc disease with up to Grade I spondylolisthesis at the target level
* Requires spinal fusion of a single level disc space (L2 to S1) with the use of local bone graft.
* Requires a posterolateral fusion procedure with or without an interbody fusion procedure using a posterior approach
* The subject has failed non-operative treatment lasting at least 6 months.

Exclusion Criteria:

* Requires spinal fusion at more than one lumbar level.
* Is pregnant, is lactating or plans to become pregnant before discontinuation of study treatment

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischgrund, MD, Principal Investigator — Corewell Health East

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted in 2 stages:
  Stage 1 was feasibility phase assessing study treatment and study assessments. LIPUS delivered via Exogen 4000+ device with a single transducer was used for this phase of the study Stage 2 was pivotal phase assessing safety and effectiveness. LIPUS delivered via Exospine device (dual transducers)
Groups:
- Exogen 4000+ Sham: Inactive LIPUS sham (single transducer)
- Exogen 4000+: Active LIPUS device (single transducer)
- Exospine: Active LIPUS device (dual transducers)
- Exospine Sham: Inactive Exospine device (dual transducers)
Period: Feasibility Stage 1
Arm/Group | Exogen 4000+ Sham | Exogen 4000+ | Exospine | Exospine Sham
Started | 8 (Stage 1: Study phase to determine the feasibility of the study treatment and assessments) | 10 (Stage 1: Study phase to determine the feasibility of the study treatment and assessments) | 0 (No subjects enrolled in Stage 1/Feasibility study) | 0 (No subjects enrolled in Stage 1/Feasibility study)
Completed | 7 | 8 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Period: Pivotal Stage 2
Arm/Group | Exogen 4000+ Sham | Exogen 4000+ | Exospine | Exospine Sham
Started | 0 (No subjects enrolled in Stage 2 pivotal study phase) | 0 (No subjects enrolled in Stage 2 pivotal study phase) | 154 (Stage 2 pivotal study phase assessed safety and effectiveness of LIPUS treatment via Exospine device) | 156 (Stage 2 pivotal study phase assessed safety and effectiveness of LIPUS treatment via Exospine device)
Completed | 0 | 0 | 52 | 51
Not Completed | 0 | 0 | 102 | 105
Not completed — Adverse Event | 0 | 0 | 6 | 11
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 13 | 14
Not completed — Physician Decision | 0 | 0 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 20 | 14
Not completed — Study Terminated by Sponsor | 0 | 0 | 60 | 63

BASELINE CHARACTERISTICS:
Population: safety: all randomized subjects trained on their device
Groups:
- Exospine Sham: Inactive LIPUS device (dual transducer)
- Exospine: Active LIPUS device (dual transducer)
- Total: Total of all reporting groups
Arm/Group | Exogen 4000+ Sham | Exogen 4000+ | Exospine Sham | Exospine | Total
Number analyzed (Participants) | 8 | 10 | 156 | 154 | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 95 | 106 | 216
  >=65 years | 2 | 1 | 61 | 48 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (11.55) | 52.4 (14.39) | 58.30 (13.90) | 56.10 (13.57) | 57.20 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 95 | 90 | 195
  Male | 5 | 3 | 61 | 64 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 13 | 15 | 31
  White | 7 | 6 | 136 | 138 | 287
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Posterolateral Fusion Success at the Treated Level
Description: Fusion success at the treated level was defined as at least 2 of 3 independent blinded radiologists agree all 3 of the following criteria were met.
  1. Confirmation of bridging bone based on computed tomography (CT) evidence of a continuous bony connection between the transverse processes on both posterolateral sides, assessed using a numeric grading scale.
  2. No evidence of motion defined as <5° angulation based on flexion and extension radiographs.
  3. No evidence of translational movement defined as <3 mm difference based on flexion and extension radiographs.
Time Frame: 12 months post treatment start
Population: Full Analysis Set (FAS): all safety subjects with at least one fully adjudicated fusion assessment at the month 12 visit of assessment
Measure: Number; unit: participants
Groups:
- Exospine Sham: Exospine Inactive: dual transducers
- Exospine Active: Exospine active: dual transducers
Arm/Group | Exospine Sham | Exospine Active
Number analyzed (Participants) | 74 | 85
participants | 25 | 28
Statistical Analysis 1: Comparison: Exospine Sham vs Exospine Active; Test type: Superiority or Other; p = 0.9905, Cochran-Mantel-Haenszel; site stratified

ADVERSE EVENTS:
Time Frame: 12 months post treatment start
Groups:
- Exogen 4000+ Sham: Stage 1 Feasibility: Exogen 4000+ sham, inactive single transducer
- Exogen 4000+: Stage 1 Feasibility: Exogen 4000+, active single transducer
- Exospine Sham: Stage 2 Pivotal: Exospine sham dual transducers
- Exospine: Stage 2 Pivotal: Exospine active dual transducers
Arm/Group | Exogen 4000+ Sham | Exogen 4000+ | Exospine Sham | Exospine
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/10 | 23/156 | 18/154
Other Adverse Events (participants affected / at risk) | 5/8 | 7/10 | 56/156 | 59/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exogen 4000+ Sham (N=8) | Exogen 4000+ (N=10) | Exospine Sham (N=156) | Exospine (N=154)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrilation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Meningocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Purulen discharge (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Failure of implant (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Stupor (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exogen 4000+ Sham (N=8) | Exogen 4000+ (N=10) | Exospine Sham (N=156) | Exospine (N=154)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 17 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 19 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 16 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 11 | 14
Paraesthesia (Nervous system disorders) | 1 | 0 | 5 | 5
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 4
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculitis (Nervous system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No